CLINICAL TRIAL: NCT01342315
Title: A Randomized, Multi-Center, Double-Blind, Vehicle-Controlled Study Evaluating the Efficacy and Safety of Product 33525 in Subjects With Tinea Cruris
Brief Title: Topical Antifungal Treatment for Tinea Cruris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-1000-01
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Tinea Cruris
Keywords: Tinea Cruris, antifungal
MeSH Terms: conditions — Tinea Cruris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Product 33525
  Interventions: Drug: 33525
- Placebo (Experimental): Product 33525 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 33525 — Daily dosing
  Arms: Active
Drug: Placebo — Daily dosing
  Arms: Placebo

SUMMARY:
To determine if a topical antifungal cream is safe and effective for the treatment of tinea cruris

ELIGIBILITY:
Inclusion Criteria:

* moderate erythema, mild scaling, and moderate pruritis

Exclusion Criteria:

* pregnancy and allergies

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving complete clearance | 3 weeks post-treatment
  Signs and Symptoms Severity Score and negative Potassium Hydroxide (KOH) and Culture

SECONDARY OUTCOMES:
Proportion of patients achieving effective treatment | 1 week Post Treatment, 2 weeks Post Treatment, and 3 weeks Post Treatment
  Clinical Cure and Mycological Cure

CONTACTS AND LOCATIONS:
Overall Officials: Ron Staugaard, Study Director — Medicis Pharmaceutical
Locations (21):
- United States (17):
  - Fremont, California
  - Los Angeles, California
  - Miami, Florida
  - Miramar, Florida
  - St. Petersburg, Florida
  - Evansville, Indiana
  - Warren, Michigan
  - Paramus, New Jersey
  - Albuquerque, New Mexico
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Goodletsville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Lynchburg, Virginia
- Belize City, Belize
- San Salvador, El Salvador
- San Pedro Sula, Honduras
- Cidra, Puerto Rico